CLINICAL TRIAL: NCT05466955
Title: Slashing Two-wheeled Accidents by Leveraging Eyecare: a Stepped-wedge Cluster Randomised Controlled Trial to Assess Impact of Spectacles on Reducing Crash and Near-crash Events Among Myopic Motorcycle Drivers in Ho Chi Minh City Vietnam
Brief Title: Slashing Two-wheeled Accidents by Leveraging Eyecare
Acronym: STABLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: L.V. Prasad Eye Institute (Other); University of Medicine and Pharmacy at Ho Chi Minh City (Other); Asia Injury Prevention Foundation (Unknown); Clearly (Other); Belfast Health and Social Care Trust (Other); Transport Development and Strategy Institute, Ministry of Transport, Vietnam (Unknown); EyeCare Foundation (Unknown)
Responsible Party: Principal Investigator, Nathan Congdon, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MHLS 22_68
Record Dates: First submitted 2022-07-11; First posted 2022-07-20 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Myopia
Keywords: crash events; near-crash events; myopia; motorcycle drivers
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: STABLE is a naturalistic driving trial with a Stepped Wedge-Cluster Randomised Trial (SW-CRT) design. The unit of randomisation in STABLE is the cluster: five universities in Ho Chi Minh City, Vietnam. The design involves random, sequential crossover of clusters from control to intervention until all clusters are exposed to the study intervention. The stepped-wedge cohort design with exchangeable correlation structure will comprise six sequences (steps) of an estimated seven myopic participants per cluster, and five clusters per sequence. The duration of each sequence is 12 weeks. Participants will not be masked to whether they are in the control or intervention period but investigators assessing study outcomes will be masked to this.
Who Masked: Investigator
Masking Description: The trial will be investigator-masked, but not participant-masked, because all participants who are eligible for eye glasses will be given them. The study's outcomes, including Crash and near Crash (CNC) events per 1,000 km, self-reported visual function (Visual Function Questionnaire (VFQ-25), and CI SRQ Crash and Injury Self report Questionnaire for all crashes, Dula Dangerous Driving Index (DDDI) will be masked from assessors.
  All care will be taken to ensure that the study team are kept masked and the trial team do not foresee conditions that will require emergency unmasking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free eye glasses for un or under-corrected myopia (Experimental): Free eyeglasses for the correction of uncorrected myopia will be provided to participants at the time of enrolment into the intervention group.
  Interventions: Device: Free eye glasses for un or under-corrected myopia
- Control-No treatment (No Intervention): Participants in the control period will not have glasses but the SW-CRT design means that all trial participants with uncorrected myopia will receive free glasses by the trials' completion, and no participant will have glasses withheld after being diagnosed with un- or under-corrected myopia.

INTERVENTIONS:
Device: Free eye glasses for un or under-corrected myopia — All participants randomised to the intervention group will be provided with free eye glasses
  Arms: Free eye glasses for un or under-corrected myopia

SUMMARY:
STABLE is a stepped-wedge cluster randomised controlled trial and its primary aim is to determine whether the provision of spectacles for the correction of myopia can reduce the average number of crash-near-crash (CNC) events among eligible motorcycle drivers in Vietnam as measured under naturalistic driving conditions with the Data Acquisition System (DAS).

STABLE is designed to assess the impact of vision correction on the safety of road users in a a Low and Middle income countries (LMIC) setting. A positive trial outcome would demonstrate the safety benefits of vision correction and would create pressure for tighter regulation of drivers' vision and the promotion of vision correction.

The study will be conducted in the peri-urban universities in Ho Chi Minh City, Vietnam and 625 students from five universities will be recruited into the trial.

Before conducting the main trial, a pilot of 35 students will be recruited to test DAS and build CNC dictionary.

Duration of the trial is 33 months from enrolment to completion of primary analysis, with 18 months for data collection.

Study participants can be both male and female motorcycle drivers aged 18 to 23 years years with at least one year of driving experience; they must use their motorcycle as their primary means of transport; drive at least 25 km per week and present with un- or under-corrected myopia that can be corrected with spectacles.

Participants with any ocular or systemic abnormality affecting vision, other than un-or under-corrected myopia will be excluded from the trial.

STABLE's primary outcome is CNC events per 1,000 km driven the DAS mounted to the motorcycles of trial participants. An interim analysis of the primary outcome will take place 9 months after data collection begins. The interim analysis will be reviewed by the trial's Data Monitoring and Ethics Committee. Unless a change is needed because of this review, the trial's primary analysis will take place 18 months after the DAS units are fitted to participants' motorcycle).

Compliance with study glasses; self-reported visual function (driving-adapted Visual Function Questionnaire-25 [VFQ-25]); Dula Dangerous Driving Index (DDDI), for all crashes; self-reported CNC events for comparison with recorded CNC events and total delivery cost per CNC event avoided with the intervention (indicator of cost-effectiveness).

DETAILED DESCRIPTION:
The primary aim of STABLE is to determine whether the provision of spectacles for the correction of myopia can reduce the average number of crash-near-crash (CNC) events among young motorcycle drivers in Vietnam.

Road traffic crashes kill more people aged 5 to 29 years worldwide than any other cause and are predicted to become the 7th leading global causes of death for all ages by 2030. The Southeast Asia has among the world's highest burdens of traffic mortality, with 20.7 fatalities per 100,000 population. The United Nations reports that motorcycles account for 93.3% of all motorized vehicles on the road in Vietnam, the highest number as a proportion of all motorized vehicles of any Association of Southeast Asian Nations country.

The investigators recently published a meta-analysis in Lancet Global Health which revealed that drivers with poor vision in Low and Middle-Income Countries (LMICs) had a 46% greater risk of experiencing a road traffic crash than those with good vision Risk Ratio (RR) 1·46, 95% Confidence Interval 1·20 to 1·78, p<0·001, 13 studies). Nevertheless, the impact of poor vision on the safety of young road users in LMICs, where many drivers do not undergo vision testing, remains poorly understood. There is a particular dearth of information for adolescent drivers, who are at greatest risk for crash-related death and the lack of reliable data has proven a significant barrier to inference of cause and effect.

Trials with robust measurement of CNC events with appropriate equipment under conditions of naturalistic driving are needed, and these have become possible only recently, due in part to falling costs and aggressive miniaturisation of GPS and on-board video systems.

STABLE will be the first cluster randomised controlled trial to investigate whether there is a link between vision correction with glasses and road safety in a LMIC.

Rationale for Intervention: The intervention in STABLE is the provision of glasses for the correction of presenting distance visual acuity <= 6/12 in the better-seeing eye due to un- or under-corrected myopia following an eye examination. The intervention will be applied to male and female motorcycle users between ages 18 and 23 enrolled at universities in Ho Chi Minh City, Vietnam

Rationale for Comparator The comparator in STABLE is standard eyecare. For university students in Vietnam, this requires the individual to pay for eyecare services provided by trained ophthalmologists or optometrists and access to good-quality eyecare services amongst university students is low. This is illustrated by the high proportion either not wearing glasses, or having glasses with incorrect power in the unpublished study noted above.

STABLE is an investigator-masked mixed-methods naturalistic driving study using a stepped-wedge cluster randomised trial (SW-CRT) design. It uses a SW-CRT design because, in a conventional parallel group cluster randomised trial, half the clusters would be randomly assigned to the intervention condition and half to the control condition. This approach would necessitate identifying participants with un- or under-corrected myopia and withholding glasses from them if they were randomly assigned to the control group until after the completion of the trial. The STABLE investigators maintain that it would be unethical to withhold glasses from motorcycle drivers who have been identified as needing them through the trial's processes for this length of time. Therefore, working with local stakeholders in Vietnam they agreed on the use of the SW-CRT design, which balances the need to conduct a randomised evaluation of the intervention with the ethical demand to provide glasses to trial participants as soon as their need for vision correction is identified.

Primary objective: is to provide reliable estimates of the impact that vision correction with glasses has on the number of CNC events in a Low- and Middle-Income Country (LMIC) setting.

Secondary objectives: are to investigate the effects of study interventions on self-reported visual function; self-reported crashes for comparison with DAS recorded crashes, and the total delivery cost per crash event avoided.

Recruitment Methods: The research team will approach the Board of Executives of the five universities and explain the purpose of the study and invite them to join the study. If they agree to participate and depending on their assignment, trial partners Asia Injury Prevention Foundation will work with each university's Department of Student Affairs and/or the Student Unions to announce, advertise and follow up on trial recruitment activities. The trial will be advertised on posters, through email and through fan page of either the Department of Student Affairs or the Student Unions.

Informed consent: to participate in STABLE will be sought from 5,200 students in 5 faculties from each university (a total of 25 clusters), to perform a self-assessment of their vision using the WHO's free smartphone-based screening app, WHOeyes. Data Acquisition System(DAS) units will be fit to the motorcycles of 625 drivers (25 per cluster), with an estimated 250 (40% of those that fail the WHOeye self-assessment) judged to be eligible for vision correction and therefore assigned to the intervention condition over the course of the trial. A 30% dropout is anticipated, yielding complete datasets from 175 trial participants.Those who meet the inclusion criteria for DAS fitting and informed consent will undergo the informed consent procedure. 35 students will be recruited from the university to be involved in the pilot study, and 175 students (35 per cluster) will be recruited from each of the other five universities for the main trial.

Sequence generation: At each sequence (step), a centralised, password-protected web-based system will be used to randomly select five clusters from those that have not yet been assigned to STABLE's intervention group. The PI on site, or an individual with delegated authority, will access the system to generate the list of five randomly selected clusters.

Diversified Technical Systems (DTS) has developed the DAS for STABLE to support the research questions and objectives of the trial. The DAS will be connected to two colour, wide-angle view video cameras: forward-facing and driver-facing. Additional data streams include: 3-axis accelerometer, Geographic Positioning System (GPS), braking and ground speed.

DAS will be fitted on site to the motorcycles of eligible students who provide informed consent to participate in the trial. For the pilot study this will take place in the week prior to the start of the pilot study. For the main trial this will take place in the month preceding the start of the trial. It will take approximately 7 days to complete DAS fitting at each university, and approximately 35 days to fit the DAS to the motorcycles of all 625 participants.

Data collection and study Instruments: Trial data collection instruments will be used to capture the outcome measures. Data collection from DAS will begin after each DAS unit has been installed on the motorcycles of consenting participants. In the main trial, the first eye examination will take place 12 weeks after the last DAS unit is fitted. After the first eye examination DAS data will only be collected from those who:

* are in a cluster that has not yet been randomly selected for transition from the control period, or
* have undergone an eye examination and been diagnosed with uncorrected myopia or under-corrected myopia (and thereby entered the intervention group) The DAS systems will be removed from the motorcycles of those participants who have had an eye examination and do not meet the inclusion criteria for assignment to the intervention group. This process will be repeated at each sequence, until DAS data are being collected from only those who meet the inclusion criteria for assignment to the intervention group (myopes only). DAS data will be collected from these DAS units up until the time they are removed from the motorcycles. Data collection from all 35 clusters will cease after the final 5 clusters in the sequence have completed 12 weeks of follow up.

Prospective participants will be contacted by email and Short Messaging Service and asked to complete a screening questionnaire to know their age, ownership of bike.

Participants who meet the inclusion criteria for DAS fitting and informed consent will be contacted again and asked to provide the following information by questionnaire:

Data Collection Data Collection

* KoboToolbox
* CRF 1 - Eligibility for Informed Consent and DAS Fitting
* CRF 2 - Baseline Assessment (VFQ 25, Dula Dangerous Driving Index)
* CRF 3 Part 1 - Before DAS Fitting
* CRF 3 Part 2 - After DAS Fitting
* CRF 5 - Vision Function Follow-up Assessment
* CRF 6 - USB Swap
* CRF 7 - Crash Report 19
* MACRO
* CRF 4 - Vision Examination
* Protocol Deviation Form
* Adverse Event Form
* Serious Adverse Event Form
* Off Study Form
* PI Sign Off Form Data will be collected using a mix of electronic and paper Case Report Forms (CRF).

Data capture by AIPF will be facilitated via KoboToolbox. Data capture by NICTU will be facilitated via MACRO.

KoboToolbox

* CRF 1 - Eligibility for Informed Consent and DAS Fitting
* CRF 2 - Baseline Assessment (VFQ 25, Dula Dangerous Driving Index)
* CRF 3 Part 1 - Before DAS Fitting
* CRF 3 Part 2 - After DAS Fitting
* CRF 5 - Vision Function Follow-up Assessment
* CRF 6 - USB Swap
* CRF 7 - Crash Report

MACRO

* CRF 4 - Vision Examination
* Protocol Deviation Form
* Adverse Event Form
* Serious Adverse Event Form
* Off Study Form
* PI Sign Off Form

Assessments in the event of a crash: Crash and Injury Self-Report Questionnaire (CI SRQ) will be collected from each participant involved in a crash event that results in hospitalisation. During the main trial, research assistants will maintain contact with participants by Short Messaging Service (SMS) on a twice monthly basis to retrieve DAS data and ensure that they are motivated to continue with the study.

Statistical Methods: Baseline demographic and clinical characteristics will be reported for all participants who are eligible for the intervention group for whom the data is available. Baseline characteristics will be summarised by means and standard deviations, medians and inter-quartile ranges, or numbers and percentages as appropriate.

Analysis of the primary outcome will use the mixed effects Poisson regression model. If the outcome includes a large number of zero values, a zero-inflated mixed effects Poisson model will be applied. In the presence of overdispersion, we will use a zero-inflated mixed effects negative binomial model. If any of these models fail to converge, a linear mixed effects model will be used as an alternative.

Null hypotheses and analyses for secondary outcomes take a similar form to that for the primary outcome. Mean differences for continuous outcomes and risk differences for binary outcomes will be reported (all adjusting for cluster, secular and time effects).

An agreement analysis will be done to compare VFQ-25 total scores at baseline and four weeks after receiving spectacles. Assuming that the response will be from the same participant and the time will be fixed, we will use the ICC and the concordance correlation coefficient (CCC) to estimate the agreement between the baseline and four weeks results.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for DAS fitting

Students from selected universities will be eligible to participate if they:

* are aged 18 to 23 years
* have at least one year or more years of driving experience
* are the sole user of their motorcycle
* use their motorcycle as their primary means of transport
* drive at least 25 km per week (self-report)
* hold a valid driving license if their motorcycle has an engine capacity >50cc

Inclusion criteria for assignment to Intervention group

Participants will be eligible for assignment to transition into the intervention group if, during the STABLE clinical examination, they are found to have:

* presenting distance visual acuity <= 6/12 in the better-seeing eye due to un- or under-corrected myopia,
* vision correctable to 6/7.5 or better in both eyes
* at least 0.5 Dioptre of myopia

Exclusion Criteria:

Individuals with any ocular or systemic abnormalities affecting vision will be ineligible to participate.

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 625 (Estimated)
Dates: Start 2024-09-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Crash and near-crash (CNC) events per 1,000 km driven | up to18 months
  CNC events as measured by Global Positioning System (GPS) and a gyroscopic sensor-video data-acquisition system (DAS) mounted to the motorcycles of trial participants.

SECONDARY OUTCOMES:
Cost-effectiveness | 18 months, Collected at the end of the trial.
  Total delivery cost per CNC event avoided with the intervention is the indicator of cost-effectiveness
Self-reported crashes | up to 18 months
  self- reported crashes compared with Data Aquisition System reported crashes and injuries are assessed using the questionnaire (Crash and Injury Self-Report Questionnaire [CI SRQ]).
Spectacle compliance | up to 18 months
  Glasses wear compliance will be assessed throughout the trial using a driver-facing camera mounted on the motorcycle's handlebars.
Visual Function | VFQ-25 is administered at baseline and one month after receiving glasses.
  Visual Function is assessed by self-reported visual function (driving-adapted Visual Function Questionnaire-25 [VFQ-25]).

CONTACTS AND LOCATIONS:
Overall Officials: Tô Gia Kiên, PhD, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City Vietnam
Locations (1):
- University of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City, Hong Bang Ward 11, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
All Individual Participant Data (IPD) will be stored in anonymised format. The IPD that includes personal identifiable information will be deleted when the data collection process is complete and before the initiation of data analysis. Only de-identified data will be shared with all the researchers for analysis.The primary analysis will be conducted on all outcome data obtained from all enrolled participants as randomised.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: All deidentified IPD will be available from February 2023 (anticipated Trial start date) to December 2025 (inclusive of analysis, publication and archival).
Access Criteria: STABLE's research team will not provide any government with direct and unfettered access to trial participant data. Government authorities seeking access to trial data must follow applicable legal processes and supply a warrant, court order for content or a subpoena for trial data.

REFERENCES:
- [Background] Peden M, Oyegbite K, Ozanne-Smith J, Hyder AA, Branche C, Rahman AKMF, Rivara F, Bartolomeos K, editors. World Report on Child Injury Prevention. Geneva: World Health Organization; 2008. Available from http://www.ncbi.nlm.nih.gov/books/NBK310641/ PMID 26269872
- [Background] Dolgin E. The myopia boom. Nature. 2015 Mar 19;519(7543):276-8. doi: 10.1038/519276a. No abstract available. PMID 25788077
- [Background] Morgan IG, French AN, Ashby RS, Guo X, Ding X, He M, Rose KA. The epidemics of myopia: Aetiology and prevention. Prog Retin Eye Res. 2018 Jan;62:134-149. doi: 10.1016/j.preteyeres.2017.09.004. Epub 2017 Sep 23. PMID 28951126
- [Background] Holden BA, Fricke TR, Wilson DA, Jong M, Naidoo KS, Sankaridurg P, Wong TY, Naduvilath TJ, Resnikoff S. Global Prevalence of Myopia and High Myopia and Temporal Trends from 2000 through 2050. Ophthalmology. 2016 May;123(5):1036-42. doi: 10.1016/j.ophtha.2016.01.006. Epub 2016 Feb 11. PMID 26875007
- [Background] Paudel P, Ramson P, Naduvilath T, Wilson D, Phuong HT, Ho SM, Giap NV. Prevalence of vision impairment and refractive error in school children in Ba Ria - Vung Tau province, Vietnam. Clin Exp Ophthalmol. 2014 Apr;42(3):217-26. doi: 10.1111/ceo.12273. Epub 2014 Jan 28. PMID 24299145
- [Background] Limburg H, Gilbert C, Hon DN, Dung NC, Hoang TH. Prevalence and causes of blindness in children in Vietnam. Ophthalmology. 2012 Feb;119(2):355-61. doi: 10.1016/j.ophtha.2011.07.037. Epub 2011 Oct 27. PMID 22035577
- [Background] Ma X, Zhou Z, Yi H, Pang X, Shi Y, Chen Q, Meltzer ME, le Cessie S, He M, Rozelle S, Liu Y, Congdon N. Effect of providing free glasses on children's educational outcomes in China: cluster randomized controlled trial. BMJ. 2014 Sep 23;349:g5740. doi: 10.1136/bmj.g5740. PMID 25249453
- [Background] Wang X, Yi H, Lu L, Zhang L, Ma X, Jin L, Zhang H, Naidoo KS, Minto H, Zou H, Rozelle S, Congdon N. Population Prevalence of Need for Spectacles and Spectacle Ownership Among Urban Migrant Children in Eastern China. JAMA Ophthalmol. 2015 Dec;133(12):1399-406. doi: 10.1001/jamaophthalmol.2015.3513. PMID 26426113
- [Background] Piyasena P, Olvera-Herrera VO, Chan VF, Clarke M, Wright DM, MacKenzie G, Virgili G, Congdon N. Vision impairment and traffic safety outcomes in low-income and middle-income countries: a systematic review and meta-analysis. Lancet Glob Health. 2021 Oct;9(10):e1411-e1422. doi: 10.1016/S2214-109X(21)00303-X. Epub 2021 Aug 16. PMID 34411516
- [Background] Pepple G, Adio A. Visual function of drivers and its relationship to road traffic accidents in Urban Africa. Springerplus. 2014 Jan 24;3:47. doi: 10.1186/2193-1801-3-47. eCollection 2014. PMID 24505558
- [Background] Swain TA, McGwin G Jr, Wood JM, Antin JF, Owsley C. Naturalistic Driving Techniques and Association of Visual Risk Factors With At-Fault Crashes and Near Crashes by Older Drivers With Vision Impairment. JAMA Ophthalmol. 2021 Jun 1;139(6):639-645. doi: 10.1001/jamaophthalmol.2021.0862. PMID 33914022
- [Background] Hanowski RJ, Hickman JS, Olson RL, Bocanegra J. Evaluating the 2003 revised hours-of-service regulations for truck drivers: the impact of time-on-task on critical incident risk. Accid Anal Prev. 2009 Mar;41(2):268-75. doi: 10.1016/j.aap.2008.11.007. Epub 2008 Dec 25. PMID 19245885
- [Background] Simons-Morton BG, Gershon P, O'Brien F, Gensler G, Klauer SG, Ehsani JP, Zhu C, Gore-Langton RE, Dingus TA. Crash rates over time among younger and older drivers in the SHRP 2 naturalistic driving study. J Safety Res. 2020 Jun;73:245-251. doi: 10.1016/j.jsr.2020.03.001. Epub 2020 Apr 8. PMID 32563399
- [Background] Klauer SG, Guo F, Simons-Morton BG, Ouimet MC, Lee SE, Dingus TA. Distracted driving and risk of road crashes among novice and experienced drivers. N Engl J Med. 2014 Jan 2;370(1):54-9. doi: 10.1056/NEJMsa1204142. PMID 24382065
- [Background] Guo F, Klauer SG, Fang Y, Hankey JM, Antin JF, Perez MA, Lee SE, Dingus TA. The effects of age on crash risk associated with driver distraction. Int J Epidemiol. 2017 Feb 1;46(1):258-265. doi: 10.1093/ije/dyw234. PMID 28338711
- [Background] Hemming K, Taljaard M. Reflection on modern methods: when is a stepped-wedge cluster randomized trial a good study design choice? Int J Epidemiol. 2020 Jun 1;49(3):1043-1052. doi: 10.1093/ije/dyaa077. PMID 32386407
- [Background] Hemming K, Taljaard M, McKenzie JE, Hooper R, Copas A, Thompson JA, Dixon-Woods M, Aldcroft A, Doussau A, Grayling M, Kristunas C, Goldstein CE, Campbell MK, Girling A, Eldridge S, Campbell MJ, Lilford RJ, Weijer C, Forbes AB, Grimshaw JM. Reporting of stepped wedge cluster randomised trials: extension of the CONSORT 2010 statement with explanation and elaboration. BMJ. 2018 Nov 9;363:k1614. doi: 10.1136/bmj.k1614. PMID 30413417
- [Background] Hemming K, Taljaard M, Grimshaw J. Introducing the new CONSORT extension for stepped-wedge cluster randomised trials. Trials. 2019 Jan 18;20(1):68. doi: 10.1186/s13063-018-3116-3. PMID 30658677
- [Background] Willemsen J, Dula CS, Declercq F, Verhaeghe P. The Dula Dangerous Driving Index: an investigation of reliability and validity across cultures. Accid Anal Prev. 2008 Mar;40(2):798-806. doi: 10.1016/j.aap.2007.09.019. Epub 2007 Oct 8. PMID 18329435
- [Background] Espie S, Boubezoul A, Aupetit S, Bouaziz S. Data collection and processing tools for naturalistic study of powered two-wheelers users' behaviours. Accid Anal Prev. 2013 Sep;58:330-9. doi: 10.1016/j.aap.2013.03.012. Epub 2013 Mar 29. PMID 23659861
- [Background] Foss RD, Goodwin AH. Distracted driver behaviors and distracting conditions among adolescent drivers: findings from a naturalistic driving study. J Adolesc Health. 2014 May;54(5 Suppl):S50-60. doi: 10.1016/j.jadohealth.2014.01.005. PMID 24759441
- [Background] Kahan BC, Morris TP. Reporting and analysis of trials using stratified randomisation in leading medical journals: review and reanalysis. BMJ. 2012 Sep 14;345:e5840. doi: 10.1136/bmj.e5840. PMID 22983531
- [Background] Permutt T. Testing for imbalance of covariates in controlled experiments. Stat Med. 1990 Dec;9(12):1455-62. doi: 10.1002/sim.4780091209. PMID 2281233
- [Background] Pocock SJ, Assmann SE, Enos LE, Kasten LE. Subgroup analysis, covariate adjustment and baseline comparisons in clinical trial reporting: current practice and problems. Stat Med. 2002 Oct 15;21(19):2917-30. doi: 10.1002/sim.1296. PMID 12325108
- [Background] Senn SJ. Covariate imbalance and random allocation in clinical trials. Stat Med. 1989 Apr;8(4):467-75. doi: 10.1002/sim.4780080410. PMID 2727470
- [Background] Sandelowski M. Whatever happened to qualitative description? Res Nurs Health. 2000 Aug;23(4):334-40. doi: 10.1002/1098-240x(200008)23:43.0.co;2-g. PMID 10940958
- [Background] Munn Z, Peters MDJ, Stern C, Tufanaru C, McArthur A, Aromataris E. Systematic review or scoping review? Guidance for authors when choosing between a systematic or scoping review approach. BMC Med Res Methodol. 2018 Nov 19;18(1):143. doi: 10.1186/s12874-018-0611-x. PMID 30453902
- [Background] Ustun TB, Chatterji S, Kostanjsek N, Rehm J, Kennedy C, Epping-Jordan J, Saxena S, von Korff M, Pull C; WHO/NIH Joint Project. Developing the World Health Organization Disability Assessment Schedule 2.0. Bull World Health Organ. 2010 Nov 1;88(11):815-23. doi: 10.2471/BLT.09.067231. Epub 2010 May 20. PMID 21076562
- [Background] Erlingsson C, Brysiewicz P. A hands-on guide to doing content analysis. Afr J Emerg Med. 2017 Sep;7(3):93-99. doi: 10.1016/j.afjem.2017.08.001. Epub 2017 Aug 21. PMID 30456117
- [Background] Guerrero-Castaneda RF, Menezes TMO, Ojeda-Vargas MG. Characteristics of the phenomenological interview in nursing research. Rev Gaucha Enferm. 2017 Jul 6;38(2):e67458. doi: 10.1590/1983-1447.2017.02.67458. English, Spanish. PMID 28700028
- [Background] Peat G, Rodriguez A, Smith J. Interpretive phenomenological analysis applied to healthcare research. Evid Based Nurs. 2019 Jan;22(1):7-9. doi: 10.1136/ebnurs-2018-103017. Epub 2018 Dec 1. No abstract available. PMID 30504450
- [Background] Akl EA, Treweek S, Foy R, Francis J, Oxman AD; ReBEQI group. NorthStar, a support tool for the design and evaluation of quality improvement interventions in healthcare. Implement Sci. 2007 Jun 26;2:19. doi: 10.1186/1748-5908-2-19. PMID 17594495
- [Background] Moore GF, Audrey S, Barker M, Bond L, Bonell C, Hardeman W, Moore L, O'Cathain A, Tinati T, Wight D, Baird J. Process evaluation of complex interventions: Medical Research Council guidance. BMJ. 2015 Mar 19;350:h1258. doi: 10.1136/bmj.h1258. PMID 25791983
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Grant A, Treweek S, Dreischulte T, Foy R, Guthrie B. Process evaluations for cluster-randomised trials of complex interventions: a proposed framework for design and reporting. Trials. 2013 Jan 12;14:15. doi: 10.1186/1745-6215-14-15. PMID 23311722
- [Background] Forero R, Nahidi S, De Costa J, Mohsin M, Fitzgerald G, Gibson N, McCarthy S, Aboagye-Sarfo P. Application of four-dimension criteria to assess rigour of qualitative research in emergency medicine. BMC Health Serv Res. 2018 Feb 17;18(1):120. doi: 10.1186/s12913-018-2915-2. PMID 29454350
- [Background] Hadi MA, Jose Closs S. Ensuring rigour and trustworthiness of qualitative research in clinical pharmacy. Int J Clin Pharm. 2016 Jun;38(3):641-6. doi: 10.1007/s11096-015-0237-6. Epub 2015 Dec 14. PMID 26666909
- [Background] Tong A, Sainsbury P, Craig J. Consolidated criteria for reporting qualitative research (COREQ): a 32-item checklist for interviews and focus groups. Int J Qual Health Care. 2007 Dec;19(6):349-57. doi: 10.1093/intqhc/mzm042. Epub 2007 Sep 14. PMID 17872937
- [Background] Tudur Smith C, Hopkins C, Sydes MR, Woolfall K, Clarke M, Murray G, Williamson P. How should individual participant data (IPD) from publicly funded clinical trials be shared? BMC Med. 2015 Dec 17;13:298. doi: 10.1186/s12916-015-0532-z. PMID 26675031
- [Background] Tudur Smith C, Nevitt S, Appelbe D, Appleton R, Dixon P, Harrison J, Marson A, Williamson P, Tremain E. Resource implications of preparing individual participant data from a clinical trial to share with external researchers. Trials. 2017 Jul 17;18(1):319. doi: 10.1186/s13063-017-2067-4. PMID 28712359
- [Background] World Health Organization. Global status report on road safety 2015. Geneva: World Health Organization; 2015
- [Background] United Nations General Assembly. Transforming our world : the 2030 Agenda for Sustainable Development: UN General Assembly; 2015
- [Background] United Nations General Assembly. Road Safety Performance Review-Vietnam. New York: United Nation; 2018.
- [Background] Hoàng Ngọc Chương HHK, Nguyễn Tịnh Anh. Assessment of freshman visual acuity and refractive error at the National Technical College of Medicine. Da Nang: University of Da Nang; 2010
- [Background] Cochrane Effective Practice and Organization of Care. EPOC Low and middle income country filters. 2020. https://epoc.cochrane.org/lmic-filters (accessed 18 March 2021)
- [Background] World Health Organization. Global status report on road safety 2018. Geneva: World Health Organization; 2018
- [Background] Ibrahim MKAMJ, H. Abdul Manan, M.M. Hanowski, R.J. Roaming the Virtual Lanes: Motorcyclists' Lane Filtering- Splitting Manoeuvres and Exposure to Road Crashes. Journal of the Society of Automotive Engineers Malaysia 2019; 3(2): 229-35
- [Background] Grove K, Soccolich S, Engström J, Hanowski R. Driver visual behavior while using adaptive cruise control on commercial motor vehicles. Transportation Research Part F: Traffic Psychology and Behaviour 2019; 60: 343-52
- [Background] Hanowski RJ. The Naturalistic Study of Distracted Driving: Moving from Research to Practice. SAE Int J Commer Veh 2011; 4(1): 286-319
- [Background] Dingus TA, Klauer SG, Neale VL, et al. The 100-Car Naturalistic Driving Study: Phase II-Results of the 100-Car Field Experiment. Report DOT HS 810 593: National Highway Traffic Safety Administration, U.S. Department of Transportation; 2006
- [Background] AAAM's Abbreviated Injury Scale.,. 2014. https://web.archive.org/web/20140328041758/http://www.aaam.org/about-ais.html (accessed 07 September 2021.
- [Background] Taplin DH, Rasic M. Facilitator's source book: Sourcebook for facilitators leading theory of change development sessions. 2012. https://www.theoryofchange.org/wp-content/uploads/toco_library/pdf/ToCFacilitatorSourcebook.pdf (accessed 01 October 2021)
- [Background] Lockwood C, Porrit K, Munn Z, et al. Systematic reviews of qualitative evidence. In: Aromataris E, Munn Z, eds. JBI Manual for Evidence Synthesis. JBI; 2020.
- [Background] Green J. Effective Sexual Health Interventions: Issues In Experimental Evaluation. Sex Transm Infect 2004; 80(1): 77-8
- [Background] Rogers EM. Diffusion of Innovations, 5th Edition. 5th ed. Riverside: Free Press; 2003
- [Background] Pawson R, Tilley N, Ebscohost. Realistic evaluation. Los Angeles: Sage; 2008
- [Background] Westhorp G. Realist impact evaluation: an introduction. London: Overseas Development Institute.,, 2014
- [Background] Shenton AK. Strategies for ensuring trustworthiness in qualitative research projects. Education for Information 2004; 22: 63-75
- [Derived] Le VC, To KG, Le VD, Nguyen L, MacKenzie G, Sigwadhi LN, Piyasena P, Tran M, Chan VF, Khanna RC, Clarke M, Lohfeld L, Dickey H, Azuara-Blanco A, Mettla AL, Rayasam S, Doan HTN, Van Do D, Le PH, Klauer C, Hanowski R, Bowden Z, Murphy L, Thompson J, McMullan S, McDowell C, Narayanan R, Little JA, Ha HT, Yoon S, Goel R, Luong L, Nguyen X, Congdon N. STABLE trial of spectacle provision and driving safety among myopic motorcycle users in Vietnam: study protocol for a stepped-wedge, cluster randomised trial. Trials. 2024 Dec 18;25(1):825. doi: 10.1186/s13063-024-08644-2. PMID 39695859